CLINICAL TRIAL: NCT03295903
Title: The Effects of Cannabinoids on Vascular and Cognitive Function in Young and Old Healthy Adults.
Brief Title: Cannabinoid Supplementation on Vascular and Cognitive Function
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Lexaria Bioscience Corp. (Industry)
Responsible Party: Principal Investigator, Phil Ainslie, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H17-01957
Record Dates: First submitted 2017-09-20; First posted 2017-09-28 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Diet Modification
Keywords: Vascular function; Cannabidiol supplementation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Sugar pill that will have no effect.
  Interventions: Dietary Supplement: Cannabidiol supplement
- Cannabidiol and herbal capsules (1 dose) (Active Comparator): Cannabidiol supplement with added ginseng, ginkgo biloba, and organic hemp oil.
  Interventions: Dietary Supplement: Cannabidiol supplement
- Cannabidiol (1 dose) (Active Comparator): Only cannabidiol supplement.
  Interventions: Dietary Supplement: Cannabidiol supplement
- Cannabidiol and herbal capsules (2 dose) (Active Comparator): Cannabidiol supplement with added ginseng, ginkgo biloba, and organic hemp oil.
  Interventions: Dietary Supplement: Cannabidiol supplement
- Cannabidiol only (2 dose) (Active Comparator): Only cannabidiol supplement.
  Interventions: Dietary Supplement: Cannabidiol supplement

INTERVENTIONS:
Dietary Supplement: Cannabidiol supplement — Subjects will be administered in a double-blinded, randomized and cross-over design

SUMMARY:
Cannabidiol (CBD) is a bioactive cannabinoid compound in marijuana (cannabis sativa), but unlike Δ9 tetrahydrocannabinol (THC), lacks the psychoactivity effect of THC. Available evidence suggests that there are marked therapeutic CBD effects for diverse disease processes including inflammation, cancers, psychosis, and epileptic seizures. The purpose of this study, in both younger and older healthy humans, is to improve our understanding of how CBD might control and regulate blood vessel health as well as cognitive and exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* non-obese
* between the ages of 18-30 & 60-75 years
* have no history of cardiopulmonary, liver, gastrointestinal, kidney or cerebrovascular disease.

Exclusion Criteria:

* are obese
* are taking prescription drugs or over-the-counter supplements that influence cardiovascular or nitric oxide metabolism
* have a history of smoking
* have history of cardiovascular, respiratory (including asthma) or neurological disease
* have known intolerance to ginseng or ginkgo herbals
* have kidney, gastrointestinal or liver disease
* have epilepsy
* have diabetes
* are pregnant or breast feeding
* do not speak English as first language
* a student in the University of British Columbia (UBC) Okanagan Centre for Heart, Lung and Vascular Health
* medical or recreational use of cannabis
* clinically diagnosed anxiety or depression
* history of opioid use
* unwilling or unable to execute the informed consent documentation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Circulating cannabidiol and nitric oxide markers | Through study completion, an average of 1 year
  Measured by venous blood sampling
Vascular function | Through study completion, an average of 1 year
  Duplex ultrasound system

SECONDARY OUTCOMES:
Height | Through study completion, an average of 1 year
  Height in cm
Weight | Through study completion, an average of 1 year
  Weight in kg
Body mass index | Through study completion, an average of 1 year
  Body mass in kilograms divided by height in meters squared
Systolic blood pressure | Through study completion, an average of 1 year
  Measured by automated sphygmomanometer
Diastolic blood pressure | Through study completion, an average of 1 year
  Measured by automated sphygmomanometer
Heart rate | Through study completion, an average of 1 year
  Measured by 3-lead electrocardiogram
Respiration | Through study completion, an average of 1 year
  Measured by spirometry
Medical History Questionnaire | Through study completion, an average of 1 year
  Assesses inclusion/exclusion criteria and prior history of medical conditions.
Gastrointestinal Distress Questionnaire | Through study completion, an average of 1 year
  Measured using a 10 cm visual analogue scale
Anxiety Questionnaire | Through study completion, an average of 1 year
  Assessed with a visual analog scale
Cognitive performance | Through study completion, an average of 1 year
  Computerized battery of neuropsychological tests
Exercise performance | Through study completion, an average of 1 year
  Step-wise exercise test on cycle ergometer

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual values will be reported in figures if applicable.

REFERENCES:
- [Derived] Patrician A, Versic-Bratincevic M, Mijacika T, Banic I, Marendic M, Sutlovic D, Dujic Z, Ainslie PN. Examination of a New Delivery Approach for Oral Cannabidiol in Healthy Subjects: A Randomized, Double-Blinded, Placebo-Controlled Pharmacokinetics Study. Adv Ther. 2019 Nov;36(11):3196-3210. doi: 10.1007/s12325-019-01074-6. Epub 2019 Sep 12. PMID 31512143